CLINICAL TRIAL: NCT03390595
Title: Phase II Multicentre, Randomized, Open-label Study to Evaluate the Safety and Efficacy of Avelumab With Gemcitabine/Carboplatin Versus Gemcitabine/Carboplatin Alone in Patients With Unresectable or Metastatic Urothelial Carcinoma (UC) Who Have Not Received Prior Systemic Therapy and Who Are Ineligible to Receive Cisplatin-based Therapy.
Brief Title: Avelumab Plus Carboplatin-gemcitabine in Urothelial Carcinoma
Acronym: INDUCOMAIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Associació per a la Recerca Oncologica, Spain (Other)
Collaborators: Merck, S.L., Spain (Industry); Pivotal S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS100070_0160; 2017-004260-36 (EudraCT Number)
Record Dates: First submitted 2017-12-21; First posted 2018-01-04 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Metastatic Urothelial Cancer
Keywords: Urothelial carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — avelumab; Carboplatin; Gemcitabine; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Avelumab plus gemcitabine/carboplatin (Experimental): 2 cycles of induction avelumab 10mg/kg every 2 weeks followed by 6 cycles of carboplatin/gemcitabine plus avelumab (carboplatin 5AUC day +1, gemcitabine 1000mg/m2 day +1 and +8 and avelumab 10mg/kg day +15) every 3 weeks followed by avelumab monotherapy 10mg/kg every 2 weeks until progressive disease or intolerance.
  Interventions: Combination Product: avelumab 10mg/kg with carboplatin/gemcitabine
- Gemcitabine/carboplatin alone (Active Comparator): patients will receive 6 cycles of carboplatin/gemcitabine (carboplatin 5AUC day +1, gemcitabine 1000mg/m2 day +1 and +8) every 3 weeks.
  Interventions: Combination Product: carboplatin/gemcitabine alone

INTERVENTIONS:
Combination Product: avelumab 10mg/kg with carboplatin/gemcitabine — Dosage and schedule:
  * Avelumab 10mg/kg will be administered over 60 minutes in the experimental arm as follows:
    * Intravenously every 2 weeks for two cycles.
    * During carboplatin-gemcitabine treatment, on day +15 (carboplatin will be administered on day 1; gemcitabine on days 1 and 8), for six cycles. Intravenously every 2 weeks until progressive disease o intolerance.
    * Intravenously every 2 weeks until progressive disease or intolerance.
  * Carboplatin-gemcitabine will be administered for six cycles, every three weeks, with the following posology, according to the SmPC
    * Carboplatin 5AUC day +1.
    * Gemcitabine 1000mg/m2 day +1 and +8.
  Other Names: Bavencio
  Arms: Avelumab plus gemcitabine/carboplatin
Combination Product: carboplatin/gemcitabine alone — •Carboplatin-gemcitabine will be administered for six cycles, every three weeks, with the following posology, according to the SmPC
  * Carboplatin 5AUC day +1.
  * Gemcitabine 1000mg/m2 day +1 and +8.
  Other Names: Standard of care for UC treatment
  Arms: Gemcitabine/carboplatin alone

SUMMARY:
Phase II Multicentre, randomized, open-label study to evaluate the safety and efficacy of avelumab with gemcitabine/carboplatin versus gemcitabine/carboplatin alone in patients with unresectable or metastatic urothelial carcinoma (UC) who have not received prior systemic therapy and who are ineligible to receive cisplatin-based therapy.

DETAILED DESCRIPTION:
The aim of this study is to evaluate if the response rates (complete response [CR] + partial response [PR]) are sufficiently high and the severe acute toxicity rates acceptably low. Patients must be cisplatin-ineligible as defined by consensus criteria (see Inclusion criteria). Patients who experience disease progression >12 months following completion of a platinum-based adjuvant or neoadjuvant regimen will also be eligible for enrolment into the study.

Once it is confirmed that the subjects fulfil the eligibility criteria and have signed the informed consent form, they will be randomized in a 1:1 ratio to receive avelumab in combination with gemcitabine/carboplatin or gemcitabine/carboplatin alone as follows:

* Arm A: patients will receive 2 cycles of induction avelumab 10mg/kg every 2 weeks followed by 6 cycles of carboplatin/gemcitabine plus avelumab (carboplatin 5AUC day +1, gemcitabine 1000mg/m2 day +1 and +8 and avelumab 10mg/kg day +15) every 3 weeks followed by avelumab monotherapy 10mg/kg every 2 weeks until progressive disease or intolerance.
* Arm B: patients will receive 6 cycles of carboplatin/gemcitabine (carboplatin 5AUC day +1, gemcitabine 1000mg/m2 day +1 and +8) every 3 weeks.

Random assignment of treatment will be stratified by the presence or absence of visceral metastasis and ECOG < 2 versus ECOG 2.

All the patients enrolled in avelumab arm will receive avelumab monotherapy maintenance until disease progression or intolerable/unacceptable toxicity. Patients in the carboplatin-gemcitabine arm, will receive up to six cycles of treatment. Tumour evaluations will be scheduled every 6 weeks (±2 weeks) during carboplatin-gemcitabine treatment (in case of cycle delay this tumour evaluations every 6 weeks should be maintained to avoid any bias in the assessment of date of progression with appropriate imaging studies for response evaluation) and every 9 weeks thereafter until progressive disease (during this period, patients at arm A will be receiving avelumab maintenance treatment).

Patients with disease progression during the treatment phase will be withdrawn from the study and will receive their treatment according to the investigator's judgment and monitored to evaluate OS.

If a patient withdraws consent and refuses to receive more treatment, the patient must be followed up for survival. If a patient withdraws consent and refuses to continue in the study, the follow-up evaluations must be discontinued.

If at the moment of end of study there would be any patient still on maintenance treatment with avelumab, Sponsor will have commitment to provide the study drug in case patient is having clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has given written informed consent stating that he or she understands the purpose of the study and the procedures involved and agrees to participate in the study.
2. The patient has histologically confirmed unresectable UC (T4b, any N; or any T, N2-3) or metastatic (M1, Stage IV) UC of the urinary tract, including renal pelvis, ureters, urinary bladder, and urethra
3. No prior systemic therapy for inoperable locally advanced or metastatic UC. For patients who received prior adjuvant/neoadjuvant chemotherapy or chemo radiation for UC, a treatment-free interval >12 months between the last treatment administration and the date of recurrence is required in order to be considered treatment naive in the metastatic setting.
4. Ineligible ("unfit") for cisplatin-based chemotherapy as defined by any one of the following criteria:

   1. Impaired renal function (GFR <60 mL/min)
   2. ECOG performance status of 2
   3. Grade ≥2 hearing loss (measured by audiometry) or ≥25 dB at two contiguous frequencies
   4. Grade ≥2 peripheral neuropathy * Criteria 4a and b are mutually exclusive: those patients with ECOG 2 won't be allowed to have an impaired renal function. For rest of the criteria, several of them may coexist.
5. The patient has at least one measurable tumour lesion (measurable disease, as defined by the RECIST criteria v1.1). If all sites of measurable disease have been irradiated, one site must have demonstrated growth after irradiation.
6. Age ≥18 years.
7. ECOG PS 0-2.
8. Life expectancy of at least 12 weeks.
9. Adequate hematologic, hepatic, and renal function, defined by:

   1. Platelet count ≥100 x10^9/L.
   2. Hemoglobin ≥ 9 g/dL (may have been transfused).
   3. Absolute neutrophil count (ANC) ≥1.5x10^9/L.
   4. Serum creatinine value not clinically significant; if creatinine >1.5 times the upper limit of normality (ULN), creatinine clearance will be calculated according to Chronic Kidney Disease Epidemiology group (CKD-EPI) formula or local formula and patients with creatinine clearance <30 mL/min shall be excluded.

      NOTE: The CKD-EPI formula for creatinine clearance is as follows:

      GFR = 141 x min(Scr/κ,1)^α x max(Scr/κ,1)^-1.209 x 0.993^Age x 1.018 [if female] x 1.159 [if black].

      Where Scr is serum creatinine (mg/dL), κ is 0.7 for females and 0.9 for males, α is -0.329 for females and -0.411 for males, min indicates the minimum of Scr/κ or 1, and max indicates the maximum of Scr/κ or 1.
   5. Alanine aminotransferase (ALT/SGPT), aspartate aminotransferase (AST/SGOT) and alkaline phosphatase (AP) ≤2.5 ×ULN (≤5 ×ULN in the presence of liver metastasis), unless this AP increase is explained due to the presence of bone metastases (with patient matching ALT, AST and bilirubin criteria), and serum total bilirubin ≤1.5 ×ULN.
10. Archival or newly-obtained representative formalin-fixed paraffin-embedded (FFPE) tumor specimens in paraffin blocks must be available.
11. Females of childbearing potential must have a negative serum pregnancy test within 7 days of study entry. Patients of childbearing potential who participate in this study must use effective contraceptive methods (e.g., abstinence, intrauterine device, oral or injectable contraceptives, a double barrier method or surgical sterility) to prevent pregnancy starting as soon as the informed consent form is signed and continuing for at least 13 weeks after the last dose of the study medication is administered.

Exclusion Criteria:

1. Women who are currently pregnant or breast-feeding.
2. Persisting toxicity related to prior therapy (NCI CTCAE v. 4.03 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable.
3. Patients who had undergone major surgery, radiation therapy or treatment with chemotherapy or any investigational agent within 28 days prior to Study day 1.
4. Evidence of severe or uncontrolled systemic disease or any concurrent condition (including uncontrolled diabetes mellitus) which in the Investigator's opinion makes it undesirable for the subject to participate in the study or which would jeopardize compliance with the protocol.
5. History of another neoplasm. However, patients with prior history of either non-metastatic non melanoma skin cancers; carcinoma in situ of the cervix; or cancer cured by surgery, small field radiation or chemotherapy ≥3 years prior to randomisation; or treated patients with early stage and low risk prostate cancer (≤pT2 N0 M0, Gleason ≤6 and Prostate-specific antigen [PSA] ≤0.5 ng/mL) at study entry will be eligible.
6. Prior allogeneic stem cell or solid organ transplantation, or active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. However, patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible
7. Current use of immunosuppressive medication, EXCEPT for the following:

   1. Intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection);
   2. Systemic corticosteroids at doses ≤10 mg/day of prednisone or equivalent;
   3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
8. History of pulmonary fibrosis.
9. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrolment), myocardial infarction (< 6 months prior to enrolment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
10. Known history of testing positive for HIV or known acquired immunodeficiency syndrome.
11. Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive).
12. Active tuberculosis.
13. Active infection requiring systemic therapy.
14. Vaccination within 4 weeks of the first dose of avelumab and while on trials is prohibited except for administration of inactivated vaccines.
15. Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v4.03 Grade ≥ 3).
16. Other severe acute or chronic medical conditions including colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behaviour; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 24 months
  The ORR is defined as the sum of the complete and partial responses (CR+PR), (according to Response Evaluation Criteria in Solid Tumours [RECIST criteria v1.1] and iRECIST).

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 24 months
  Time from randomisation to either documented disease progression or death from any cause (whichever occurs earlier).
Overall Survival (OS) | 24 months
  Time from randomisation to death from any cause. Patients still alive at the time of OS analysis will be censored on their last date of contact. Patients who withdraw from the study without having completed the withdrawal consent will be followed up to determine their status whenever possible.
  For the purposes of this study, subjects should be evaluated every 6 weeks with the appropriate imaging technique according to each centre's routine practice, during the combined treatment, and every 9 weeks during the maintenance period. In case of cycle delay every 6 weeks should be maintained to avoid any bias in the assessment of the date of progression with the appropriate imaging studies for response evaluation. Response will be monitored as per the RECIST 1.1 criteria.
Duration of Response (DoR) | 24 months
  Time from the first confirmation of objective response according to RECIST 1.1 criteria until disease progression or death.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 24 months
  Incidence and severity of adverse events. AEs will be coded and evaluated using the National Cancer Institute, Common Toxicity criteria for Adverse Events (NCI-CTCAE) v4.03 toxicity criteria (if NCI-CTCAE are not applicable, the Medical Dictionary for Regulatory Activities [MedDRA] will be used).

OTHER OUTCOMES:
Analysis of pathologic resistance mechanisms to treatment combination | 24 months
  Determination of resistance mechanisms in disease's biopsies, describing the pathologic features that may predict response or resistance to treatment.
Analysis of immunologic resistance mechanisms to treatment combination | 24 months
  Determination of resistance mechanisms in blood serum, describing the immunologic features that may predict response or resistance to treatment.
Analysis of genomic resistance mechanisms to treatment combination | 24 months
  Determination of PD-L1 expression in tumor infiltrating immune cells and in tumor cells (pre and post-treatment samples will be analyzed).

CONTACTS AND LOCATIONS:
Overall Officials: Joaquín Bellmunt, MD, PhD, Principal Investigator — Hospital del Mar; Alejo Rodríguez-Vida, MD, PhD, Principal Investigator — Hospital del Mar
Locations (15):
- Spain (15):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Instituto Catalán de Oncología (ICO L'Hospitalet) - H. Durán i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Fundación Althaia - Xarxa Assistencial Univ. de Manresa, Manresa, Barcelona
  - Hospital Universitario Parc Tauli, Sabadell, Barcelona
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital del Mar, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clìnic de Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Universitario Virgen del Rocío, Seville
  - Fundación Instituto Valenciano de Oncología, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bajorin DF, Dodd PM, Mazumdar M, Fazzari M, McCaffrey JA, Scher HI, Herr H, Higgins G, Boyle MG. Long-term survival in metastatic transitional-cell carcinoma and prognostic factors predicting outcome of therapy. J Clin Oncol. 1999 Oct;17(10):3173-81. doi: 10.1200/JCO.1999.17.10.3173. PMID 10506615
- [Background] Ferlay J, Shin HR, Bray F, Forman D, Mathers C, Parkin DM. Estimates of worldwide burden of cancer in 2008: GLOBOCAN 2008. Int J Cancer. 2010 Dec 15;127(12):2893-917. doi: 10.1002/ijc.25516. PMID 21351269
- [Background] Ferlay J, Parkin DM, Steliarova-Foucher E. Estimates of cancer incidence and mortality in Europe in 2008. Eur J Cancer. 2010 Mar;46(4):765-81. doi: 10.1016/j.ejca.2009.12.014. Epub 2010 Jan 29. PMID 20116997
- [Background] Witjes JA, Comperat E, Cowan NC, De Santis M, Gakis G, Lebret T, Ribal MJ, Van der Heijden AG, Sherif A; European Association of Urology. EAU guidelines on muscle-invasive and metastatic bladder cancer: summary of the 2013 guidelines. Eur Urol. 2014 Apr;65(4):778-92. doi: 10.1016/j.eururo.2013.11.046. Epub 2013 Dec 12. PMID 24373477
- [Background] AJCC cancer staging manual. 7th ed. New York: Springer, pp. 497-502.
- [Background] National Comprehensive Cancer Network (2011) NCCN clinical practice guidelines for bladder cancer. www nccn org.
- [Background] Bellmunt J, Albiol S. New chemotherapy combinations for advanced bladder cancer. Curr Opin Urol. 2001 Sep;11(5):517-22. doi: 10.1097/00042307-200109000-00011. PMID 11493774
- [Background] Loehrer PJ Sr, Einhorn LH, Elson PJ, Crawford ED, Kuebler P, Tannock I, Raghavan D, Stuart-Harris R, Sarosdy MF, Lowe BA, et al. A randomized comparison of cisplatin alone or in combination with methotrexate, vinblastine, and doxorubicin in patients with metastatic urothelial carcinoma: a cooperative group study. J Clin Oncol. 1992 Jul;10(7):1066-73. doi: 10.1200/JCO.1992.10.7.1066. PMID 1607913
- [Background] Galsky MD, Hahn NM, Rosenberg J, Sonpavde G, Hutson T, Oh WK, Dreicer R, Vogelzang N, Sternberg CN, Bajorin DF, Bellmunt J. Treatment of patients with metastatic urothelial cancer "unfit" for Cisplatin-based chemotherapy. J Clin Oncol. 2011 Jun 10;29(17):2432-8. doi: 10.1200/JCO.2011.34.8433. Epub 2011 May 9. PMID 21555688
- [Background] De Santis M, Bellmunt J, Mead G, Kerst JM, Leahy M, Maroto P, Gil T, Marreaud S, Daugaard G, Skoneczna I, Collette S, Lorent J, de Wit R, Sylvester R. Randomized phase II/III trial assessing gemcitabine/carboplatin and methotrexate/carboplatin/vinblastine in patients with advanced urothelial cancer who are unfit for cisplatin-based chemotherapy: EORTC study 30986. J Clin Oncol. 2012 Jan 10;30(2):191-9. doi: 10.1200/JCO.2011.37.3571. Epub 2011 Dec 12. PMID 22162575
- [Background] Dogliotti L, Carteni G, Siena S, Bertetto O, Martoni A, Bono A, Amadori D, Onat H, Marini L. Gemcitabine plus cisplatin versus gemcitabine plus carboplatin as first-line chemotherapy in advanced transitional cell carcinoma of the urothelium: results of a randomized phase 2 trial. Eur Urol. 2007 Jul;52(1):134-41. doi: 10.1016/j.eururo.2006.12.029. Epub 2006 Dec 26. PMID 17207911
- [Background] Rosenberg JE, Hoffman-Censits J, Powles T, van der Heijden MS, Balar AV, Necchi A, Dawson N, O'Donnell PH, Balmanoukian A, Loriot Y, Srinivas S, Retz MM, Grivas P, Joseph RW, Galsky MD, Fleming MT, Petrylak DP, Perez-Gracia JL, Burris HA, Castellano D, Canil C, Bellmunt J, Bajorin D, Nickles D, Bourgon R, Frampton GM, Cui N, Mariathasan S, Abidoye O, Fine GD, Dreicer R. Atezolizumab in patients with locally advanced and metastatic urothelial carcinoma who have progressed following treatment with platinum-based chemotherapy: a single-arm, multicentre, phase 2 trial. Lancet. 2016 May 7;387(10031):1909-20. doi: 10.1016/S0140-6736(16)00561-4. Epub 2016 Mar 4. PMID 26952546
- [Background] Plimack ER, et al. Pembrolizumab (MK-3475) for advanced urothelial cancer: Updated results and biomarker analysis from KEYNOTE-012. J Clin Oncol 33, 2015 (suppl;abstr 4502).
- [Background] Massard C, Gordon MS, Sharma S, Rafii S, Wainberg ZA, Luke J, Curiel TJ, Colon-Otero G, Hamid O, Sanborn RE, O'Donnell PH, Drakaki A, Tan W, Kurland JF, Rebelatto MC, Jin X, Blake-Haskins JA, Gupta A, Segal NH. Safety and Efficacy of Durvalumab (MEDI4736), an Anti-Programmed Cell Death Ligand-1 Immune Checkpoint Inhibitor, in Patients With Advanced Urothelial Bladder Cancer. J Clin Oncol. 2016 Sep 10;34(26):3119-25. doi: 10.1200/JCO.2016.67.9761. Epub 2016 Jun 6. PMID 27269937
- [Background] Galsky M, et al. Efficacy and safety of nivolumab monotherapy in patients with metastatic urothelial cancer (mUC) who have received prior treatment: Results from the phase II CheckMate 275 study. Presented at ESMO 2016 (abstract LBA31_PR).
- [Background] http://www.mercknewsroom.com/news-release/oncology-newsroom/mercks-keynote-045-studying-keytruda-pembrolizumab-advanced-bladder-c.
- [Background] Balar AV, Galsky MD, Rosenberg JE, Powles T, Petrylak DP, Bellmunt J, Loriot Y, Necchi A, Hoffman-Censits J, Perez-Gracia JL, Dawson NA, van der Heijden MS, Dreicer R, Srinivas S, Retz MM, Joseph RW, Drakaki A, Vaishampayan UN, Sridhar SS, Quinn DI, Duran I, Shaffer DR, Eigl BJ, Grivas PD, Yu EY, Li S, Kadel EE 3rd, Boyd Z, Bourgon R, Hegde PS, Mariathasan S, Thastrom A, Abidoye OO, Fine GD, Bajorin DF; IMvigor210 Study Group. Atezolizumab as first-line treatment in cisplatin-ineligible patients with locally advanced and metastatic urothelial carcinoma: a single-arm, multicentre, phase 2 trial. Lancet. 2017 Jan 7;389(10064):67-76. doi: 10.1016/S0140-6736(16)32455-2. Epub 2016 Dec 8. PMID 27939400
- [Background] Balar A, et al. Pembrolizumab (pembro) as first-line therapy for advanced/unresectable or metastatic urothelial cancer: Preliminary results from the phase 2 KEYNOTE-052 study. Presented at ESMO 2016 (abstract LBA32_PR).
- [Background] Patel M. R., Ellerton J. A., Infante J. R., et al. Avelumab in patients with metastatic urothelial carcinoma: pooled results from two cohorts of the phase 1b JAVELIN solid tumor trial. Journal of Clinical Oncology. 2017;35(supplement 6S) doi: 10.1200/JCO.2017.35.6_suppl.330. abstract 330.
- [Background] Apolo AB, Infante JR, Balmanoukian A, Patel MR, Wang D, Kelly K, Mega AE, Britten CD, Ravaud A, Mita AC, Safran H, Stinchcombe TE, Srdanov M, Gelb AB, Schlichting M, Chin K, Gulley JL. Avelumab, an Anti-Programmed Death-Ligand 1 Antibody, In Patients With Refractory Metastatic Urothelial Carcinoma: Results From a Multicenter, Phase Ib Study. J Clin Oncol. 2017 Jul 1;35(19):2117-2124. doi: 10.1200/JCO.2016.71.6795. Epub 2017 Apr 4. PMID 28375787
- [Background] Heery CR, O'Sullivan-Coyne G, Madan RA, Cordes L, Rajan A, Rauckhorst M, Lamping E, Oyelakin I, Marte JL, Lepone LM, Donahue RN, Grenga I, Cuillerot JM, Neuteboom B, Heydebreck AV, Chin K, Schlom J, Gulley JL. Avelumab for metastatic or locally advanced previously treated solid tumours (JAVELIN Solid Tumor): a phase 1a, multicohort, dose-escalation trial. Lancet Oncol. 2017 May;18(5):587-598. doi: 10.1016/S1470-2045(17)30239-5. Epub 2017 Mar 31. PMID 28373007
- [Background] Bracci L, Schiavoni G, Sistigu A, Belardelli F. Immune-based mechanisms of cytotoxic chemotherapy: implications for the design of novel and rationale-based combined treatments against cancer. Cell Death Differ. 2014 Jan;21(1):15-25. doi: 10.1038/cdd.2013.67. Epub 2013 Jun 21. PMID 23787994
- [Background] Lynch TJ, Bondarenko I, Luft A, Serwatowski P, Barlesi F, Chacko R, Sebastian M, Neal J, Lu H, Cuillerot JM, Reck M. Ipilimumab in combination with paclitaxel and carboplatin as first-line treatment in stage IIIB/IV non-small-cell lung cancer: results from a randomized, double-blind, multicenter phase II study. J Clin Oncol. 2012 Jun 10;30(17):2046-54. doi: 10.1200/JCO.2011.38.4032. Epub 2012 Apr 30. PMID 22547592
- [Background] Reck M, Bondarenko I, Luft A, Serwatowski P, Barlesi F, Chacko R, Sebastian M, Lu H, Cuillerot JM, Lynch TJ. Ipilimumab in combination with paclitaxel and carboplatin as first-line therapy in extensive-disease-small-cell lung cancer: results from a randomized, double-blind, multicenter phase 2 trial. Ann Oncol. 2013 Jan;24(1):75-83. doi: 10.1093/annonc/mds213. Epub 2012 Aug 2. PMID 22858559
- [Background] Hamilton G, Rath B. Avelumab: combining immune checkpoint inhibition and antibody-dependent cytotoxicity. Expert Opin Biol Ther. 2017 Apr;17(4):515-523. doi: 10.1080/14712598.2017.1294156. Epub 2017 Feb 22. PMID 28274143
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- [Background] Rodriguez-Vida A, Bellmunt J. Avelumab for the treatment of urothelial cancer. Expert Rev Anticancer Ther. 2018 May;18(5):421-429. doi: 10.1080/14737140.2018.1448271. Epub 2018 Mar 14. PMID 29540084
- [Background] Rodriguez Vida A et al. Phase II randomized study of first line avelumab with carboplatin-gemcitabine versus carboplatin-gemcitabine alone in patients with metastatic urothelial carcinoma ineligible for cisplatin-based therapy. DOI: 10.1200/JCO.2018.36.15_suppl.TPS4591 Journal of Clinical Oncology 36, no. 15_suppl.
- [Result] Perez Valderrama B et al. LBA27 - Phase II multicenter, randomized study to evaluate efficacy and safety of avelumab with gemcitabine/carboplatin (CG) vs CG alone in patients with unresectable or metastatic urothelial carcinoma (mUC) who are ineligible to receive cisplatin-based therapy. Annals of Oncology (2020) 31 (suppl_4): S1142-S1215. 10.1016/annonc/annonc325.
- See also: APRO Website — https://apro.es/